CLINICAL TRIAL: NCT06760052
Title: Longitudinal Data Registry of a Spectrum of Plasma Cell Dyscrasia with Long-term Follow-up
Brief Title: Longitudinal Data Registry of Plasma Cell Dyscrasia
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Peng Liu, Zhongshan Hospital, Fudan University, Shanghai Zhongshan Hospital
Other Study IDs: SHZS-PCD-001
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Multiple Myeloma and Other Plasma Cell Neoplasms
MeSH Terms: conditions — Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Enrolled patients: The final personalized management strategy is determined based on both current conventional treatment options and physicians' and patients' preferences. The following agents might be applied: proteasome inhibitors (PIs), immunomodulatory drugs (IMiDs), alkylating agents, anti-CD38 monoclonal antibodies, bispecific antibodies, and cell therapy, with or without steroids.

SUMMARY:
This study aims to identify clinical characteristics, response and clinical outcome of plasma cell dyscrasia (PCD) diagnosed in Zhongshan Hospital, Fudan University from May 2023. In its current version, the registry incorporates historical data (collected from 2007) and is prospectively collecting follow-up data and recording patient outcomes.

DETAILED DESCRIPTION:
PCD is a spectrum of diseases that is being gradually understood in Asia. This study aims to observe and describe the clinical and genetic characteristics of Chinese PCD patients, and to explore the relationship between the characteristics and pathogenesis. It also aims to discover the potential distinct clonal evolution patterns among different subtype of this disease spectrum. This study is a non-interventional real-world, study. Alll registered data are collected from real clinical practice cases. The medical data includes patient demographic, tumor characteristics, laboratory examination, history of treatments, adverse reactions, efficacy results and possible prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

Patients with pathological diagnosis of PCD [e.g.: symptomatic/asymptomatic multiple myeloma, monoclonal gammopathy of undetermined significance (MGUS), POEMS syndrome, light chain (AL) amyloidosis) from 2007 to 2027 in Zhonshan Hospital.

Patients who had complete diagnostic, treatment and follow-up records. With fully comprehension and signature of the informed consent form (ICF) for participation.

Exclusion Criteria:

Patients who refused to use reliable methods of contraception during pregnancy, lactation or age-appropriate period.

Patients who suffered from severe mental illness. Patients who were deemed unsuitable for inclusion by the investigator.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pathological diagnosis of PCD from 2007 to 2027 according to 2016 WHO classification.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the time of enrollment to data cut-off (Up to approximately 20 years).
  Overall survival (OS) refers to the time from receiving the first dose of regimen to death of any cause.

SECONDARY OUTCOMES:
Progression-free survival | From the time of enrollment to data cut-off (Up to approximately 20 years).
  Progression-free survival (PFS) is defined as the time from the date of first administration to the date of first disease progression or death of any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No